CLINICAL TRIAL: NCT06921915
Title: Viewing Woman-Centered, Animated, Explainer Videos From the Confident Bladder Website to Optimize Bladder Health and Toileting Management Behaviors: A Randomized Controlled Trial in Community-Based Women at Midlife
Brief Title: Efficacy of Animated Videos to Foster Healthy Bladder Behaviors in Community Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kathleen O'Connell (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor-Investigator, Kathleen O'Connell, Isabel Maitland Stewart Professor of Nursing Education Emerita, Teachers College, Columbia University
Organization: Teachers College, Columbia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 24-305
Record Dates: First submitted 2024-08-26; First posted 2025-04-10 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2024-08

CONDITIONS: Urinary Bladder, Overactive; Urinary Incontinence, Urge
Keywords: Prevention; Learning; Clinical trials, randomized
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This online study administered by Qualtrics Research Services randomly allocates study participants to groups. The participants don't know which group until they are assigned after they complete surveys. The group assignments are masked for the investigators and outcomes assessor until after data collection is completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- eLearning Daytime (Experimental): This group completes pre-intervention surveys and then is assigned to view the part of the website that deals with Daytime Hold Confidence. Participants engage in an elearning activity on how to prevent and deal with urinary urges during daytime activities. Participants in the group complete post-intervention surveys immediately after viewing the website and two weeks after study entry.
  Interventions: Other: eLearning
- eLearning Sleep/Wake (Experimental): This group completes pre-intervention surveys and then is assigned to view the part of the website that deals with Sleep/Wake Confidence. Participants engage in an elearning activity on how to prevent and deal with urinary urges that occur after the participant has fallen asleep and then when they arise in the morning. In addition, this group is assigned to the Tips and Tricks, which covers additional information. Participants in the group complete post-intervention surveys immediately after viewing the website and two weeks after study entry.
  Interventions: Other: eLearning
- Control Group (No Intervention): This group completes pre-intervention surveys and then immediately completes the post-intervention surveys. Two weeks after study entry they complete the same surveys completed by members of the other two groups.

INTERVENTIONS:
Other: eLearning — Participants in the intervention arms view a website developed by urinary bladder experts that presents information about how to prevent inconvenient urinary urges.
  Other Names: eLearning Daytime
  Arms: eLearning Daytime; eLearning Sleep/Wake

SUMMARY:
In daily life, women are exposed to a wide range of challenging situations that can negatively affect toileting management and long-term bladder health. Research shows that women engage in behaviors that may lead to unfavorable consequences, such as a worrying sense of bladder urgency or an awkward moment of urine leakage. The investigators surmise that consciously or unconsciously adopted behaviors influence lifelong bladder health, toileting management, and sense of self-efficacy in this arena. Adoption of research-supported behaviors that foster bladder well-being for women is dependent on women's access to learning multiple healthy behavioral strategies.

Studies on personal woman-centered strategies for toileting management and adoption of behaviors that foster bladder health are scarce in the scientific literature. The investigators have published encouraging results of an in-person study with a clinical sample using accessible and enjoyable videos about research-based bladder health behaviors, invented by the co-investigator of this study, Janis M. Miller.

We now launch an additional study of 90 community-based women of midlife age using an online survey methodology that incorporates sending study participants to the website. The study has two main objectives:

1. To determine baseline bladder health and toileting management behavior profiles in intervention-naïve community-based women as assessed by the Confident Bladder Behavior Questionnaire
2. To determine at post-intervention whether behavioral profiles of the respondents have significantly changed after being randomized into one of three groups: Group 1: who watch the animated explainer videos within the Confident Bladder website that are predominantly related to daytime conditions, Group 2: who watch the Confident Bladder website's animated explainer videos predominantly related to sleep/wake conditions and the additional tips and tricks section, and Group 3: controls who only receive access to the the Confident Bladder website at study's end after post-intervention assessments.

We will test the following hypothesis:

Viewing the Confident Bladder website will demonstrate an effect size at 2-weeks post intervention of greater than 0.5, as determined by comparing number and percentage of research-based behavioral strategies used by the Control group to the number and percentage of strategies used by the two intervention groups who were assigned to view different parts of the website.

ELIGIBILITY:
Inclusion Criteria:

* Must have a U.S. IP Address
* Must be female between age of 40 and 64
* Must be enrolled in a Study Participant Panel accessed by Qualtrics
* Must read and speak English

Exclusion Criteria:

* NonEnglish speakers/readers
* Does not consent to participate
* Does not commit to providing thoughtful and honest answers to the surveys

Ages: 40 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2024-08-27 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2024-10-06 (Actual)

PRIMARY OUTCOMES:
The Confident Bladder Behavior Questionnaire | All respondents complete this questionnaire during the first session and then two weeks later. Respondents in the experimental arms complete the questionnaire prior to the eLearning activity.
  A 31-item questionnaire assessing the extent to which respondents engage in behaviors related to maintaining a healthy bladder.

SECONDARY OUTCOMES:
Knowledge about Healthy Bladder Behaviors | All respondents complete this test during the first study session. Those in the experimental arms complete it after they view the website.
  A 14-item multiple choice test on the information conveyed in the website.
Urinary Cues Questionnaire | All respondents complete this in the first study session and two weeks after the eLearning activity.. Those in the experimental arm complete the Urinary Cues Questionnaire before the eLearning activity.
  A 21-item survey assessing the extent to which participants recognize that each cue gives them the urge to urinate.
Self-efficacy for Performing Healthy Bladder Behaviors | All respondents complete this in the first study session and two weeks after the eLearning activity.. Those in the experimental arm complete the Self-efficacy Questionnaire after the eLearning activity.
  a 12-item survey assessing the respondents' confidence that they can carry out healthy bladder behaviors.
Evaluation of the Website and the Study | All respondents complete the Evaluation surveys during the first session only. Those in the Experimental groups complete the Evaluation survey after viewing the website.
  For Experimental groups, a 14-item questionnaire assessing the respondents' experience with the website and their intention to follow the advice offered by the website.
  For Control Group, a 4-item questionnaire assessing the respondents' experience with the study and their intention to view the Confident Bladder website after the study.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen A O'Connell, PhD, Principal Investigator — Teachers College Columbia Universit
Locations (1):
- Teachers College, Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller JM, Hawthorne KM, Park L, Tolbert M, Bies K, Garcia C, Misiunas R, Newhouse W, Smith AR. Self-Perceived Improvement in Bladder Health After Viewing a Novel Tutorial on Knack Use: A Randomized Controlled Trial Pilot Study. J Womens Health (Larchmt). 2020 Oct;29(10):1319-1327. doi: 10.1089/jwh.2018.7606. Epub 2019 Dec 3. PMID 31800360